CLINICAL TRIAL: NCT01021982
Title: Objective Perimetry in Normal Subjects,Glaucoma Patients and Retinitis Pigmentosa Patients .
Brief Title: Evaluation of Objective Perimetry Using Pupillometer
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University, Claire and Amedee Maratier Institute (Unknown)
Responsible Party: Principal Investigator, Dr. Ygal Rotenstreich, Director, Electrophysiology Clinic, Goldschleger Eye Institute, Sheba Medical Center
Other Study IDs: SHEBA-09-6958-AS-CTIL
Record Dates: First submitted 2009-11-29; First posted 2009-12-01 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Retinitis Pigmentosa; Glaucoma; Visual Field
Keywords: Pupillometer; Retinitis Pigmentosa; Glaucoma; Objective perimetry
MeSH Terms: conditions — Retinitis Pigmentosa; Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Glaucoma: Glaucoma Patients with visual field defects
- Retinitis Pigmentosa: Retinitis Pigmentosa Patients with visual field defects

SUMMARY:
Objective perimetry can better monitor visual field defects in RP and Glaucoma patients than conventional subjective perimetry.The PLR ( Pupil Light Reflex ) of the short and long wave ratio should be significantly higher in areas of visual field defects in RP and Glaucoma patients.

DETAILED DESCRIPTION:
Pupil light reflex will be measured by a pupillometer in response to short and long wavelength light small spot stimulus in different area of the visual field. The PRL will be measured in four quadrant, central, 10, 20, and 30 degree from the visual axis.

Stimulus duration will be 1000 ms (1 sec), with intervals of 890 ms between stimuli. The stimuli size V with light intensity of 39.8 cd-s/m2 for both short wavelength stimuli (peak 485 nm) and long wavelength stimuli (peak 620nm).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75
2. Sign on informed consent
3. Papillary response to light.
4. Groups of : Normal , Glaucoma patients with early glaucoma damage on HVF (nasal step ect. ), Glaucoma patients with advanced glaucoma damage on HVF (arcuate , tubular vision ) and RP patients (Early VF damage , ring scotoma ) .
5. Refractive correction up to -3.5 D.

Exclusion Criteria:

1. Cloudy corneas.
2. Surgical intraocular ophthalmic procedure within the past 30 days.
3. Nonreactive pupils.
4. Synechia of the iris to the lens after surgery or inflammation .
5. Neovascularization.
6. Iris coloboma.
7. Sphincter damage due to ischemia or trauma (tears of sphincter or diffuse damage to muscle).
8. Sphincter damage due to high intraocular pressure .
9. Iris tumor or cyst .
10. Ectropion uvea .
11. Adie's pupil .
12. Optic neuropathy with the potential for producing a positive RAPD (Relative Afferent Pupillary Defect ).
13. Chronic use of myotics or mydriatics.
14. Systemic Medication which affect on papillary response .
15. Any condition preventing accurate measurement or examination of the pupils.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
PLR response amplitude and latency | Not defined yet

CONTACTS AND LOCATIONS:
Overall Officials: Ygal Rotenstreich, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel, Israel

REFERENCES:
- [Background] Yoshitomi T, Matsui T, Tanakadate A, Ishikawa S. Comparison of threshold visual perimetry and objective pupil perimetry in clinical patients. J Neuroophthalmol. 1999 Jun;19(2):89-99. PMID 10380129
- [Background] Kalaboukhova L, Fridhammar V, Lindblom B. Relative afferent pupillary defect in glaucoma: a pupillometric study. Acta Ophthalmol Scand. 2007 Aug;85(5):519-25. doi: 10.1111/j.1600-0420.2006.00863.x. Epub 2007 Jun 15. PMID 17573859
- [Background] Kardon RH. Pupil perimetry. Curr Opin Ophthalmol. 1992 Oct;3(5):565-70. doi: 10.1097/00055735-199210000-00002. PMID 10147922
- [Background] Kardon RH, Kirkali PA, Thompson HS. Automated pupil perimetry. Pupil field mapping in patients and normal subjects. Ophthalmology. 1991 Apr;98(4):485-95; discussion 495-6. doi: 10.1016/s0161-6420(91)32267-x. PMID 2052302
- [Derived] Skaat A, Sher I, Kolker A, Elyasiv S, Rosenfeld E, Mhajna M, Melamed S, Belkin M, Rotenstreich Y. Pupillometer-based objective chromatic perimetry in normal eyes and patients with retinal photoreceptor dystrophies. Invest Ophthalmol Vis Sci. 2013 Apr 17;54(4):2761-70. doi: 10.1167/iovs.12-11127. PMID 23482470